CLINICAL TRIAL: NCT06215872
Title: Investigation of the Effectiveness of Structured Myofacial Chain Exercise Training Applied in the Early Period After Distal Radius Fracture
Brief Title: Effectiveness of Structured Myofacial Chain Exercises After Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Atlas University (Other)
Responsible Party: Principal Investigator, Sebnem Nur Alkan, PHD Student, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAU-ALKAN-001
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Distal Radius Fractures
Keywords: Tele-Health; Exercise; Physical Therapy And Rehabilitation; Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Control Single-Blind Study
Who Masked: Participant
Masking Description: Knowledge that which exercises are structured for research will keep from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper Extremity Exercises Group (Active Comparator): Participants will treated exercises with focused on upper extremity especially wrist muscles.
  Interventions: Other: Therapeutic Exercises
- Myofascial Chains Exercises Group (Experimental): Participants will treated exercises with focused on whole body especilly myofascial chains.
  Interventions: Other: Therapeutic Exercises
- Control Group (No Intervention): Participants will do any exercises. They will join only assessment sessions.

INTERVENTIONS:
Other: Therapeutic Exercises — Participants who have inclusion criterias after DRF reconstrontion pos-op 4. week will included this study. Certified Physiotherapist who have master of science degree and doctorate student will assessed them before and after treatment with face to face. Also exercise education will give face to face with same therapist. After that first sessions patients will progress their standardize or structered exercises pragram with telerehabilition during 4 weeks and 16 sessions. All sessions will be supervised with physiotherapist. End of study assessments will perform again with same therapist.
  Arms: Myofascial Chains Exercises Group; Upper Extremity Exercises Group

SUMMARY:
When determining the treatment method to be applied in distal radius fracture (DRF), in addition to clinical and radiological evaluation, the patient's age, physical activity level, cognitive status, severity of trauma, mechanism of injury and type of fracture are important factors in the treatment plan. Clinical studies show that physiotherapy is useful in improving the limitation of movement and pain in DRF. It shows that the active movement level is increased by decreasing the level. Rehabilitation after surgery proceeds similarly to conservative treatment. When exercise approaches in the literature are examined, it is seen that specific exercises for the wrist and forearm are recommended for treatment, but it has been reported that there are not enough studies to constitute evidence value. For decades, the skeletal muscles of the human body have been characterized as independent structures. However, recent research supports the "single muscle theory", contrary to this classical view. According to this theory, the fascia tissue that covers the entire body connects the muscles to each other in the form of chains, and the muscles in the chain work together in performing functional movements. These chains are called myofascial chains. Fascia tissue that creates all these connections; It consists of tightly arranged connective tissue and is structurally similar to tendons and ligaments. It surrounds organs, muscles, vessels and nerves, connects tissues and allows them to slide and move over each other. Past histological studies have reported that there are also contractile cells in the fascia structure. Although there are problems in rehabilitation after DRF that go beyond a single segment and affect the whole body; There is no study in the literature that uses the myofascial chain exercises approach in the treatment of these problems. In the light of all this information, the thesis study aims to ensure the active participation of the upper body muscles in the rehabilitation process with the DRUK program planned with myofascial chain exercises and in this way to improve the functional level obtained as a result of rehabilitation.

DETAILED DESCRIPTION:
Clinical studies show that physiotherapy is useful in improving the limitation of movement in distal radius fractures and increases the level of active movement by reducing the level of pain. Providing functional restoration with physiotherapy not only increases the quality of life but also reduces the number of days patients cannot go to work. Rehabilitation after surgery proceeds similarly to conservative treatment. When exercise approaches in the literature are examined, it is seen that specific exercises for the wrist and forearm are recommended for treatment, but it has been reported that there are not enough studies to constitute evidence value. Due to the increased risk of prolonged immobilization and damaged tissues after surgery compared to closed reduction; If problems such as disuse atrophy, loss of proprioception and joint range of motion are taken into consideration, all upper extremity disorders may occur after surgery, including the elbow and shoulder joints, which are positioned together with the wrist and whose use is restricted. The following have been reported as early and late complications after surgical treatments: i)Complex regional pain syndrome, reflex sympathetic dystrophy, algodystrophy, compartment syndrome; ii) Tendon adhesion or rupture; iii)Nerve compression; iv) Post traumatic arthritis; v)Dupuytren's contracture. Although some of these complications are related to surgery, other complications are affected by processes involving the fascial system. For decades, the skeletal muscles of the human body have been characterized as independent structures. However, recent research supports the "single muscle theory", contrary to this classical view. According to this theory, the fascia tissue that covers the entire body connects the muscles to each other in the form of chains, and the muscles in the chain work together in performing functional movements. These chains are called myofascial chains. In cadaveric studies, mechanical force transfer along these connections has been demonstrated, and this connection has been tried to be explained with biotensegrite models. Due to this load transfer, all structures on the chain are affected by the forces or disorders that any structure in the myofascial chain is exposed to, and this is explained by the biotensivity theory. Fascia tissue that creates all these connections; It consists of tightly arranged connective tissue and is structurally similar to tendons and ligaments. It surrounds organs, muscles, vessels and nerves, connects tissues and allows them to slide and move over each other. Past histological studies have reported that there are also contractile cells in the fascia structure. Although there are problems in rehabilitation after distal radius fracture that go beyond a single segment and affect the whole body; There is no study in the literature that uses the myofascial chain exercises approach in the treatment of these problems. In the light of all this information, the thesis study aims to ensure the active participation of the upper body muscles in the rehabilitation process with the distal radius fracture program planned with myofascial chain exercises and in this way to improve the functional level obtained as a result of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-70
* Being able to establish written and verbal communication in Turkish
* Post-Op rehabilitation after primary DRF surgery, at 4 weeks, post op at 6 weeks at the l latest
* Fixation using volar plating and nailing method
* Post-op, if instruments were left temporarily, these instruments should be removed before the study
* No previous history of surgery involving the upper extremity
* To have sufficient technological device usage skills and fast internet infrastructure to use video communication technologies without any problems
* Having a device that provides the necessary equipment for video calling
* Having a table and 6 m2 of space to allow exercise in the living area

Exclusion Criteria:

* Occurrence of one of the complex regional pain syndrome subtypes after fracture
* History of any chronic systemic, rheumatological, neurological, vascular disease
* History of traumatic injury to intact extremities and trunk in the last 6 months
* Presence of pain complaints including spine and shoulder pain over 3 according to the Visual Analogue Scale
* Those who use anti-inflammatory drugs
* Presence of cognitive or psychological illness that will prevent cooperation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Quick DASH (The Disabilities of the Arm, Shoulder and Hand) | Pre treatment and end of study (4 weeks after from first assessment)
  Quick-DASH is an 11-item questionnaire that questions a person's limitations in upper extremity problems.

SECONDARY OUTCOMES:
The Visual Analogue Scale (VAS) | Pre treatment and end of study (4 weeks after from first assessment)
  This scale scores from 0 to 10. Higher scores indicate worse pain.
Hand Functional Index (HFI) | Pre treatment and end of study (4 weeks after from first assessment)
  The hand functional index scale consists of 9 items. Each item is scored between 0-3. It is calculated by adding the scores from all items separately for both hands.
Michigan Hand Outcomes Questionnaire (MHQ) | Pre treatment and end of study (4 weeks after from first assessment)
  It is a survey that includes six subheadings from patients (pain, hand function, satisfaction with hand function, work performance, ADL and aesthetic satisfaction).
Joint Range of Motion Measurement Test With Goniometer | Pre treatment and end of study (4 weeks after from first assessment)
  Joint range of motion evaluation was made with a goniometer device and flexion, extension, radial-ulnar deviation angles were evaluated.
Hand Grip Strength Measurement Test With Hand Dynamometer | Pre treatment and end of study (4 weeks after from first assessment)
  During the test, the patient was in a sitting position and the force value was recorded by squeezing the device in the palm of the hand and not supporting the body with the elbow.
Pinch Grip Strength With Pinch Meter | Pre treatment and end of study (4 weeks after from first assessment)
  The force value was recorded by the researcher, by holding the device from the indicator part and asking the subject to squeeze it between the thumb and index finger in a sitting position.
Fingertip Dexterity and Gross Movement of the Hand With The Purdue Pegboard Test (PPT) | Pre treatment and end of study (4 weeks after from first assessment)
  With materials such as metal pipe beads and sequin beads inside the device; The subject was asked to perform the exercises against the clock in the order and ways specified in the guide.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No